CLINICAL TRIAL: NCT02277509
Title: Chinese Diabetes Prevention Program: An Implementation and Dissemination Study
Brief Title: Chinese Diabetes Prevention Program (Chinese DPP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: New York Presbyterian Hospital (Other); Chinese American Independent Practice Association (CAIPA) (Other); City University of New York (Other); Pace University (Other)
Responsible Party: Principal Investigator, Judith Wylie-Rosett, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2014-3252
Record Dates: First submitted 2014-10-15; First posted 2014-10-29 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese DPP (Experimental): Our Chinese DPP intervention includes: 1) skills development core adapted from the DPP core curriculum, 2) stress reduction counseling and activities, 3) physical activity sessions, 4) self-monitoring tools for diet and physical activity, 5) barriers assessment linked to tool box, and 6) post-core support intervention.
  Interventions: Behavioral: Chinese DPP
- Minimal Intervention Control (Active Comparator): The minimal control intervention will consist of providing patients with publically available materials on diabetes prevention, which are produced in Chinese.
  Interventions: Behavioral: Minimal Intervention Control

INTERVENTIONS:
Behavioral: Chinese DPP — The Chinese DPP intervention will include core curriculum, stress reduction, physical activity sessions, and self-monitor diet and physical activity.
  .
  Other Names: Culturally adapted DPP curriculum
  Arms: Chinese DPP
Behavioral: Minimal Intervention Control — Patients will receive printed diabetes prevention materials in Chinese. Materials will be from primary from the National Diabetes Education Program and from the New York City Department off Health and Mental Hygiene. Patients will receive an educational packet at randomization and quarterly thereafter.
  Other Names: control
  Arms: Minimal Intervention Control

SUMMARY:
This study is being conducted in two phases. The first phase was a pilot implementation of the study protocol, which provided preliminary data from seeking funding for a larger scale trial. The study focused on testing the effects of a Diabetes Prevention Program (DPP) that has been adapted culturally and linguistically to address diabetes prevention among Chinese immigrants. Study implementation involves a variety capacity building community partnership initiatives. Partnering organizations within New York City (NYC) have included the Chinese Community Partnership for Health (CCPH) of New York Presbyterian Hospital of Lower Manhattan Hospital, the Chinese American Independent Practice Association (CAIPA), the Diabetes Research and Training Center of Albert Einstein College of Medicine (Einstein), and the City University of New York (CUNY) School of Public Health. More recently, our collaboration has expanded the potential for wider dissemination in collaboration with the Pace University Confucius Center of the Confucius Institute. By supporting Chinese language and cultural programs, the Confucius Institute facilitates communication with the 2 billion native Chinese speakers as migration and trade increase interactions globally.

DETAILED DESCRIPTION:
The pilot testing (Einstein Institutional Review Board Protocol #2010-491) demonstrated the acceptability and feasibility of implementing the culturally and linguistically Chinese DPP lifestyle protocol. The pilot study found that the intervention resulted in a significant weight loss and trends for glycemic (HbA1c) improvement among Chinese immigrants with prediabetes. The planned R01 funded study will address larger scale implementation to inform wider spread dissemination within the United States and globally. Our specific aims are to:

Aim 1. Evaluate the clinical effectiveness of the implementation model in a cluster randomized trial. Primary endpoints will include changes in weight and glycemia (HbA1c ) one year after randomization. Secondary endpoint will include cardiovascular risk markers, lifestyle (dietary intake and physical activity) and self-reported quality of life.

Aim 2. Evaluate the study generalizability using the RE-AIM (reach, efficacy/effectiveness, adoption, implementation and maintenance) framework. The specific evaluation questions include:

Reach: How many of the eligible patients enrolled? How representative are the study participants of the underlying population?

Efficacy/Effectiveness: How did the intervention affect participants' outcome measures?

Adoption: How acceptable were the intervention components to the participants?

Implementation: How many of the intervention components were provided as planned?

Maintenance: How much of the 1-year intervention effects are sustainable at 2-year follow-up? What mechanisms are available for sustaining the intervention?

Aim 3. Evaluate the cost-effectiveness of the implementation model with respects to weight and glycemic (HbA1c) change.

Aim 4. Disseminate "lessons learned" and effective program components to expand access to effective programs within the United States via the registry developed by the Centers for Disease Control of DPP intervention sites and to explore global dissemination issues via our partnership with Confucius Institute.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes (A1c -5.5-6.4%),
* BMI ≥ 23 kg/m2,
* ability to read and understand Chinese,
* enrollment in CAIPA network,
* ability and willingness to provide informed consent.

Exclusion Criteria:

* Diagnosis of diabetes,
* health conditions for which the lifestyle would be contra-indicated,
* inability to provide informed,
* BMI < 23 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent Change in Weight | 12 months
Percent Change in BMI | 12 months

SECONDARY OUTCOMES:
Percent HbA1c reduction | 12 months
Changes in Blood Pressure | 12 months
  Cardiovascular risk biomarkers
Changes in Lipid Profile | 12 months
  Cardiovascular risk biomarkers
Sustained changes in weight | 24 months
Sustained changes in HbA1c | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wylie-Rosett, EdD, RD, Principal Investigator — Professor, Epidemiology & Population Health
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States